CLINICAL TRIAL: NCT04538014
Title: Interventional, Open-label, Positron Emission Tomography (PET) Study With [11C]-Lu AF88434 Investigating Blood-brain Barrier Penetration, Safety, and Tolerability of Lu AF88434 in Healthy Men
Brief Title: A Study in Healthy Men to Investigate Uptake and Distribution of Lu AF88434 in the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18426A
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF88434 (Experimental)
  Interventions: Drug: Lu AF88434; Drug: [11C]-Lu AF88434

INTERVENTIONS:
Drug: Lu AF88434 — Oral solution
Drug: [11C]-Lu AF88434 — [11C]-Lu AF88434, and a radioactive dose not exceeding 400 MBq at each PET examination, intravenous bolus injection

SUMMARY:
This study will investigate how much of Lu AF88434 will get into the blood and the brain in healthy men

DETAILED DESCRIPTION:
The study consists of the following parts:

* a Screening Visit
* an MRI scanning visit
* an in-clinic stay which includes: a Safety Baseline one day prior to dosing, a one-day [11C]-Lu AF88434 imaging session consisting of a baseline PET measurement and a post-dose PET measurement conducted after the administration of a single oral dose of Lu AF88434, pharmacokinetic (PK) sampling and safety assessments throughout the period
* a Follow-up Visit 7 days after dosing

ELIGIBILITY:
Inclusion Criteria:

* The subject has a BMI ≥18.5 and ≤30.0 kg/m2 at the Screening Visit and at the Baseline Visit
* The subject has a normal MRI performed during the screening period, as judged by the investigator
* The subject is, in the opinion of the investigator, generally healthy based on the assessment of medical history, physical examination, vital signs, body weight, ECG, and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests
* The subject can tolerate confined spaces for prolonged periods of time
* The subject is suitable for radial artery blood sampling and cannulation

Exclusion Criteria:

* The subject has any concurrent disorder that may affect the particular target or absorption, distribution, or elimination of the Investigational Medicinal Product (IMP)

Other in- or exclusion criteria may apply

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Total distribution volume (VT) of [11C]-Lu AF88434 | At baseline and post-dose on Day 1
  Whole-brain distribution volume
C(PET) of Lu AF88434 | Day 1
  Mean plasma concentration of Lu AF88434 during the post-dose PET measurement
Area Under Curve (AUC(0-inf)) of Lu AF88434 | Day 1
  Area under the plasma concentration time curve of Lu AF88434 from zero to infinity
Cmax of Lu AF88434 | Day 1
  Maximum observed plasma concentration of Lu AF88434

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Parexel International Northwick Park Hospital (Level 7), Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided